CLINICAL TRIAL: NCT06411808
Title: The Impact of Sensory-Adapted Dental Environment on Anxiety and Behavior in Children With Sensory Processing Disorders: A Crossover Randomized Control Trial
Brief Title: Evaluating Sensory-Adapted Dental Care in Children With Sensory Processing Disorders
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: STUDY00000573
Record Dates: First submitted 2024-05-06; First posted 2024-05-13 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Sensory Processing Disorder
Keywords: sensory processing disorders; pediatric dentistry; dental anxiety; behavioral outcomes; sensory adaptation; crossover randomized controlled trial; sensory modulation disorder; sensory over-responsivity

STUDY DESIGN:
Intervention Model Description: Participants will receive dental care in both a standard and a sensory-adapted dental environment in a randomized order to compare effects on anxiety and behavior.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants and study personnel involved in the delivery and assessment of the treatment outcomes are blinded to the phase order to maintain the integrity of the study results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SADE Group: Sensory-Adapted Dental Environment (Experimental): Participants in this arm will experience dental care in a Sensory-Adapted Dental Environment. Modifications such as dimmed lighting, noise-canceling headphones, and specialized dental tools are used to minimize sensory overload and enhance comfort during dental procedures.
  Interventions: Behavioral: Sensory-Adapted Dental Environment
- Control Group: Regular Dental Environment (No Intervention): Participants in this arm will receive dental care in a Regular Dental Environment without sensory adaptations, representing standard dental care settings.

INTERVENTIONS:
Behavioral: Sensory-Adapted Dental Environment — The Sensory-Adapted Dental Environment (SADE) involves altering the dental setting to reduce sensory stimuli that can cause discomfort or anxiety in children with sensory processing disorders. This includes the use of controlled lighting, ambient sounds, and non-threatening tools to create a calming atmosphere conducive to positive dental experiences.
  Other Names: SADE
  Arms: SADE Group: Sensory-Adapted Dental Environment

SUMMARY:
This clinical trial examines the efficacy of a Sensory-Adapted Dental Environment (SADE) in reducing anxiety and improving behavioral outcomes in children with sensory processing disorders during routine dental visits. By modifying the dental setting to accommodate sensory sensitivities-such as using dim lighting, noise-canceling headphones, and non-threatening dental tools-the study aims to create a more comfortable dental experience for these children. This research could potentially inform broader pediatric dentistry practices, making dental care more accessible and less distressing for children with sensory sensitivities.

DETAILED DESCRIPTION:
The study is a crossover randomized controlled trial designed to assess the impact of a Sensory-Adapted Dental Environment (SADE) on children with sensory processing disorders, focusing on both physiological and behavioral responses. Participants will undergo two dental cleaning visits; one in a standard dental environment and one in a sensory-adapted setting. Each visit will be spaced three to four months apart to monitor short-term effects and behaviors. The primary outcomes measured will include changes in anxiety levels, as assessed by physiological markers (e.g., heart rate) and behavioral scales (e.g., modified dental anxiety scale). Secondary outcomes will evaluate the overall acceptance of the sensory-adapted environment by children and their caregivers. This study seeks to demonstrate that tailored environmental modifications can significantly improve the dental care experience, potentially leading to enhanced long-term dental health and reduced care avoidance among children with sensory processing disorders. The trial will also gather qualitative feedback from participants and their parents to better understand individual experiences and refine future adaptations in pediatric dental practices.

ELIGIBILITY:
Inclusion Criteria:

* Ability of subject (or Legally Authorized Representative (LAR)) to understand and the willingness to sign a written informed consent document.
* For children, informed assent and parental informed consent to participate in the study.
* Males and females; Age <5-17 years>
* Self-reported or documented diagnosis of sensory processing disorder (SPD), sensory modulation disorder (SMD), or sensory over-responsivity (SOR) based on medical records or occupational therapy evaluation. Diagnosis codes per ICD-10 may include, but are not limited to, F88 and F89 for SPD, as these are often used for atypical neurodevelopmental conditions where specific sensory challenges are present.
* A score above the threshold on the Sensory Profile-2, which indicates significant sensory processing issues.
* A history of at least one previous dental cleaning, to ensure familiarity with the dental care process.
* Willingness and ability to adhere to the study intervention regimen, including attending two dental sessions in different environmental settings (RDE and SADE).
* Ability to attend intervention sessions at the designated site, UT Health School of Dentistry.
* Access to transportation or necessary resources for participating in the study sessions at the UT Health School of Dentistry.
* Not currently undergoing orthodontic braces treatment or using anticholinergic medication, as per the exclusion criteria.

Exclusion Criteria:

* Significant developmental disabilities or medical conditions that preclude the safe conduct of dental procedures or the ability to consent, even with a Legally Authorized Representative (LAR), such as uncontrolled epilepsy or severe behavioral disorders that could lead to self-harm or harm to staff within a dental setting.
* Complex dental needs that require specialized procedures or surgeries not provided within the study's dental care setting, such as advanced orthodontic work or oral surgery, which might interfere with the study's assessments or outcomes.
* Previous traumatic dental experiences resulting in extreme dental care avoidance, as this could confound the effects of the SADE versus RDE environments.
* Current or scheduled orthodontic braces treatment during the study period, as braces may affect the child's sensory experience and response to the dental environment.
* Use of anticholinergic medication, due to their potential to alter physiological measures of stress and anxiety, which are key outcomes for this study.
* Any condition that, in the opinion of the investigators, may pose a risk to the participant's safety or may affect the study outcomes.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2024-06-28 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Effect of SADE on Heart Rate | Baseline to approximately 50 minutes (after dental appointment)
  This measure evaluates the impact of the Sensory-Adapted Dental Environment (SADE) on physiological indicators of anxiety, specifically heart rate change.
Effect of SADE on Oxygen Saturation | Baseline to approximately 50 minutes (after dental appointment)
  This measure evaluates the impact of the Sensory-Adapted Dental Environment (SADE) on physiological indicators of anxiety, specifically oxygen saturation change.
Effect of SADE on Systolic and Diastolic Blood Pressure | Baseline to approximately 50 minutes (after dental appointment)
  This measure evaluates the impact of the Sensory-Adapted Dental Environment (SADE) on physiological indicators of anxiety, with change in systolic or diastolic blood pressure.
Frankl Behavior Rating Scale Change | Baseline to approximately 50 minutes (after dental appointment)
  A change in score on the Frankl behavioral rating scale. This is a scored as a single rating of behavior between 1 and 4 with a higher score indicating a more positive attitude.
Ohio State University Behavior Rating Scale | Baseline to approximately 50 minutes (after dental appointment)
  This scale rates the participants' behavior. A change in score on the behavioral rating scale. This is a scored as a single rating of behavior between 1 and 4 with a lower score indicating a more positive attitude.
Venham's Clinical Anxiety Scale | Baseline to approximately 50 minutes (after dental appointment)
  A scale used to measure the change in clinical anxiety of participants will be a single item scored from 0-3, where a higher score indicates more anxiety and protest from the participant.
Wong Bakers Visual FACES Scale Modified | Visit 1 Day 1 to Visit 2 (May occur Day 90-120)
  A modification of Wong-Baker scale designed to understand the child's anxiety on the same scale and faces pattern, pre-visit and post-visit.

CONTACTS AND LOCATIONS:
Overall Officials: Nida-e-Haque Mahmud, DDS, BDS, Principal Investigator — UT Health San Antonio
Locations (1):
- UT Health San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share individual participant data (IPD) that underlie the results reported in this trial after de-identification. Data sets will include all collected IPD encompassing demographic, physiological, behavioral, and self-reported anxiety metrics. The shared data will support further research on sensory processing disorders and dental anxiety, enhancing the reproducibility of our results and enabling secondary analyses by other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD and supporting documentation will become available starting 6 months after the publication of the main results and remain accessible for a period of 5 years. This allows sufficient time for the research community to propose, prepare, and conduct secondary analyses.
Access Criteria: Access to the shared IPD will be granted to researchers who provide a methodologically sound proposal. Applications for access will be reviewed by an independent review committee appointed by the University of Texas Health Science Center. Criteria for evaluation will include the scientific merit of the research proposal, the research team's expertise, and the potential to contribute to scientific understanding or clinical improvement.

REFERENCES:
- [Background] Cermak SA, Stein Duker LI, Williams ME, Dawson ME, Lane CJ, Polido JC. Sensory Adapted Dental Environments to Enhance Oral Care for Children with Autism Spectrum Disorders: A Randomized Controlled Pilot Study. J Autism Dev Disord. 2015 Sep;45(9):2876-88. doi: 10.1007/s10803-015-2450-5. PMID 25931290
- [Background] Fallea A, Zuccarello R, Roccella M, Quatrosi G, Donadio S, Vetri L, Cali F. Sensory-Adapted Dental Environment for the Treatment of Patients with Autism Spectrum Disorder. Children (Basel). 2022 Mar 10;9(3):393. doi: 10.3390/children9030393. PMID 35327765
- [Background] Stein Duker LI, Como DH, Jolette C, Vigen C, Gong CL, Williams ME, Polido JC, Florindez-Cox LI, Cermak SA. Sensory Adaptations to Improve Physiological and Behavioral Distress During Dental Visits in Autistic Children: A Randomized Crossover Trial. JAMA Netw Open. 2023 Jun 1;6(6):e2316346. doi: 10.1001/jamanetworkopen.2023.16346. PMID 37266941
- [Background] Reynolds K, Chandio N, Chimoriya R, Arora A. The Effectiveness of Sensory Adaptive Dental Environments to Reduce Corresponding Negative Behaviours and Psychophysiology Responses in Children and Young People with Intellectual and Developmental Disabilities: A Protocol of a Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2022 Oct 22;19(21):13758. doi: 10.3390/ijerph192113758. PMID 36360634
- [Background] Cermak SA, Stein Duker LI, Williams ME, Lane CJ, Dawson ME, Borreson AE, Polido JC. Feasibility of a sensory-adapted dental environment for children with autism. Am J Occup Ther. 2015 May-Jun;69(3):6903220020p1-10. doi: 10.5014/ajot.2015.013714. PMID 25871593
- [Background] P BJ. Dental subscale of children's fear survey schedule and dental caries prevalence. Eur J Dent. 2013 Apr;7(2):181-185. doi: 10.4103/1305-7456.110166. PMID 24883023
- [Background] Kim G, Carrico C, Ivey C, Wunsch PB. Impact of sensory adapted dental environment on children with developmental disabilities. Spec Care Dentist. 2019 Mar;39(2):180-187. doi: 10.1111/scd.12360. Epub 2019 Feb 6. PMID 30729554
- [Background] Ismail AF, Tengku Azmi TMA, Malek WMSWA, Mallineni SK. The effect of multisensory-adapted dental environment on children's behavior toward dental treatment: A systematic review. J Indian Soc Pedod Prev Dent. 2021 Jan-Mar;39(1):2-8. doi: 10.4103/jisppd.jisppd_36_21. PMID 33885380